CLINICAL TRIAL: NCT06221683
Title: A Multicenter Clinical Study of Molecular Subtyping Combined With MRD-driven Remission Induction Regimen in Children and Adolescents With AML: A Phase II Cohort Study (GMCAII)
Brief Title: Clinical Study of Induction Therapy Options Based on Molecular Subtyping and MRD in Children and Adolescents With AML
Acronym: GMCAII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Shaoyan Hu, Study Chair, Children's Hospital of Soochow University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GMCAII
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: AML, Childhood; Acute Myeloid Leukemia
Keywords: AML; Childhood; Molecular subtyping; MRD
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Homoharringtonine; Cytarabine; Etoposide; venetoclax; Idarubicin; Sorafenib; gilteritinib; avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDC group (Experimental): Patients with CBF fusion gene (RUNX1: : RUNX1T1 and CBFB: : MYH11) or KMT2A: : MLLT3(AF9) , KMT2A: : MLLT10(AF10) , KMT2A: : MLLT4(AF6) fusion gene or KIT mutation will receive SDC regimen, including one course of HAE (Homoharringtonine, cytarabine, etoposide) in induction I. These patients will continue on the SDC (HAE) regimen in the second course if the MRD is < 1% after induction I, otherwise venetoclax will be added to the SDC group sequentially on Day 2 after the end of HAE. FLT3-ITD will be given sorafenib or gilteritinib as early as possible, and patients with KIT mutations will be recommended to add avapritinib as appropriate. These targeted drugs will not be combined with venetoclax.
  Interventions: Drug: Homoharringtonine; Drug: Cytarabine; Drug: Etoposide; Drug: Venetoclax; Drug: Sorafenib; Drug: Gilteritinib; Drug: Avapritinib
- LDC group (Experimental): Patients with the exception of the CBF fusion gene (RUNX1: : RUNX1T1 and CBFB: : MYH11) or those with the KMT2A: : MLLT3(AF9) , KMT2A: : MLLT10(AF10) , KMT2A: : MLLT4(AF6) fusion gene or KIT mutation will receive the LDC (MAG/IDAG+ venetoclax) regimen in induction I. Patients with MRD ≥1% or KIT mutations, assessed after induction I, will receive the HAE plus venetoclax (or targeted drugs) regimen, otherwise, they will receive MAG/IDAG + venetoclax. FLT3-ITD will be given sorafenib or gilteritinib as early as possible, and patients with KIT mutations will be recommended to add avapritinib as appropriate. These targeted drugs will not be combined with venetoclax.
  Interventions: Drug: Cytarabine; Drug: Mitoxantrone hydrochloride liposome; Drug: Recombinant Human Granulocyte Colony-Stimulating Factor; Drug: Idarubicin Hydrochloride; Drug: Sorafenib; Drug: Gilteritinib; Drug: Avapritinib

INTERVENTIONS:
Drug: Homoharringtonine — 3mg/m2/day for weighing >10kg, 0.1mg/kg/day for weighing ≤10kg, d1-7, ivgtt, qd, more than 6 hours
  Other Names: Homoharringtonine injection
  Arms: SDC group
Drug: Cytarabine — 100mg/m2/q12h for weighing >10kg, 3.3mg/kg/q12h for weighing ≤10kg, d1-7, ivgtt, q12h, more than 30 minutes in SDC group; 10mg/m2/q12h for weighing >10kg, 0.33mg/kg/q12h for weighing ≤10kg, d1-10, s.c.,q12h (the first dose at 8 am) in the LDC group;
  Other Names: Cytosar
Drug: Etoposide — 100mg/m2/d for weighing >10kg, 3.3mg/kg/d for weighing ≤ 10kg, d1-5, ivgtt, qd, more than 4 hours
  Other Names: Etoposide injection
  Arms: SDC group
Drug: Venetoclax — 100mg/m2/d for weighing >10kg, 3.33mg/kg/d for weighing ≤10kg, d12-25, po, qd
  Other Names: Venclexta
  Arms: SDC group
Drug: Mitoxantrone hydrochloride liposome — 5mg/m2/d for weighing >10kg, 0.17mg/kg/d for weighing ≤ 10kg, d1, 3, 5, ivgtt, qod, more than 2 hours at 10 am.
  Other Names: Mitoxantrone hydrochloride liposome injection
  Arms: LDC group
Drug: Recombinant Human Granulocyte Colony-Stimulating Factor — 5ug/kg/d, d1-10, s.c., qd, at 1pm
  Other Names: Recombinant Human Granulocyte Colony-Stimulating Factor Injection
  Arms: LDC group
Drug: Idarubicin Hydrochloride — 3mg/m2/day for weighing >10kg, 0.1mg/kg/day for weighing ≤ 10kg, d1-7, ivgtt, qd, more than 6 hours.
  Other Names: Idarubicin hydrochloride injection
  Arms: LDC group
Drug: Sorafenib — 100mg/m2/day for weighing >10kg, 3.3mg/kg/day for weighing ≤10kg, from identification, po, qd
  Other Names: Nexavar
Drug: Gilteritinib — 20mg/m2/day for weighing >10kg, 0.7mg/kg/day for weighing ≤ 10kg, from identification, po, qd
  Other Names: Xospata Pill
Drug: Avapritinib — 50mg/m2/day for weighing bodyweight >10kg, 1.65mg/kg/day for weighing ≤ 10kg, po, qd
  Other Names: AYVAKIT

SUMMARY:
The goal of this clinical trial is to estimate the rate (probability) of complete remission or complete remission with incomplete count recovery (CR/CRi) with negative MRD after induction I and II, event-free survival (EFS), and cumulative incidence (probability) of relapse (CIR), in patients receiving molecular/precision medicine and MRD-driven remission inductions, and to assess secondarily if there is an improvement over the AML2018 protocol.

DETAILED DESCRIPTION:
Advances in risk stratification and therapy, have improved the event-free survival (EFS) and overall survival (OS) for pediatric acute myeloid leukemia (AML) with current treatment strategies. Investigators previously conducted a multicenter, randomized controlled trial (AML18) to compare the efficacy and safety of low-dose chemotherapy versus standard-dose chemotherapy. The results showed that low-dose chemotherapy was non-inferior to standard-dose chemotherapy in terms of efficacy and had fewer adverse events. However, different subtypes exhibited varying treatment responses to both chemotherapy regimens. The MRD (Measurable Residual Disease) after induction therapy in both groups had an impact on prognosis. According to the backbone of the 2018 protocol, investigators decide whether to use low-dose or standard-dose for the first induction according to the patient's fusion gene, and the second induction and subsequent treatment are adjusted according to the treatment response. Patients with the following 5 fusion genes RUNX1: RUNX1T1, CBFβ: MYH11, KMT2A: MLLT3 (AF9), KMT2A: MLLT10 (AF10), KMT2A: MLLT4 (AF6) fusion or KIT mutation will be assigned to the standard dose remission induction regimen (HHT + Ara-C + VP16), others will be assigned to the standard dose regimen (Mitoxantrone/Idarubicin + Ara-C + G-CSF). At the same time, investigators will add targeted drugs such as venetoclax, avaptitinib, and gilteritinib/sorafenib to the chemotherapy regimen and assess their safety and efficacy. Post-induction consolidation consisted of 3 to 4 cycles of standard-dose chemotherapy according to risk classification. Patients classified as high-risk are candidates for allogeneic bone marrow transplantation after 1 or 2 courses of consolidation.

ELIGIBILITY:
Inclusion Criteria:

* 1、Newly diagnosed, untreated AML；
* 2、Under 18 years old;
* 3、Patients who have used hydroxyurea or cytarabine before diagnosis, but the dosage of cytarabine does not exceed 5 days, and the total dose does not exceed 500 mg/m2 (50 mg/m2, q12h × 5d)；
* 4、 Liver function：Tbil≤2×ULN, ALT/AST≤3×ULN, creatinine clearance ≥50ml/min；Cardiac NYHA grading<3；SaO2>92%;
* 5、No active infection (symptoms resolved for more than 3 days if infected)
* 6、ECOG<2;
* 7、Expected survival time greater than 12 weeks;
* 9、Obtain the consent of the child and/or guardian and sign the informed consent form.

Exclusion Criteria:

* 1、Acute megakaryocytic leukemia (AMKL)；
* 2、Acute promyelocytic leukemia (APL);
* 3、Treatment-related secondary AML and AML with definite MDS transformation；
* 4、Myeloproliferative neoplasm (such as Juvenile myelomonocytic leukemia, JMML);
* 5、AML secondary to congenital bone marrow failure (such as AML secondary to Fanconi anemia (FA)；
* 6、AML secondary to Down syndrome;
* 7、Only temporary chemotherapy, radiotherapy, or immunotherapy, but not systematic treatment according to the treatment plan;
* 8、 Temporary chemotherapy, radiotherapy, or immunotherapy only, not systemic therapy per protocol;
* 9、Having any significant abnormal concurrent disease or mental illness that impacts the life safety and compliance of the patient and impacts informed consent, study participation, follow-up, or interpretation of results. In this case, all the participating units are required to report directly to the responsible person for this project to jointly decide whether they meet the exclusion criteria；
* 10、Patients with very poor nutritional status, severe infection, cardiac insufficiency, and intolerance to chemotherapy;
* 11、Relapsed AML at any time；
* 12、The attending physician considers that the patient is not suitable for entering the study protocol based on the patient's physical condition, economic status, and other factors.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Rate of CR/CRi with negative MRD | Day 26 (HAE group) and Day 32 (MAG+Ven group) for remission induction 1 and 2 are the necessary time points for response evaluation.
  CR/CRi with negative MRD was defined as less than 5% blasts in bone marrow and MRD <0.1%.
Event-free survival | From date of treatment until the date of the occurrence of the event, whichever comes first, assessed up to 72 months. Patients remaining event-free are censored at the last follow-up time.
  Events/failures of EFS include any-cause death, relapse, second malignancy, no CR after Indiction II and off-therapy due to abandonment or attending physician's decision.
  Induction II and off-therapy due to abandonment or attending physician's decision.
Cumulative incidence of relapse | From date of treatment until the date of when a failure of CIR occurs, whichever comes first, assessed up to 72 months.
  Failures of CIR only include relapse and no CR after Induction 2. Other failures including death in resission (before repalse), second malignancy, and off-therapy due to abandonment or attending physician's decision are considered competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyan Hu, MD, PhD, Study Chair — Children 's Hospital of Soochow University
Locations (13):
- China (13):
  - First Affiliated Hospital Of University of Science and Technology of China, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Guangzhou Women and Children Medical Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Kaifeng Children's Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - XiangYa Hospital Central South University, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Children's Hospital, Xuzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Children's Hospital Of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Institute of Genomics, Chinese Academy of Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No